CLINICAL TRIAL: NCT04492696
Title: Comparison of Concussion Education Programs and Intent to Report Concussion in High School Football Athletes
Brief Title: Comparison of Concussion Education Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Shelley Goldman, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 40500
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crashcourse (Active Comparator): CC uses an approach to providing concussion education informed by user-centered formative design research studies. The program features an interactive "choose your own adventure" approach to navigate the learner through the content, and is guided by near-peer Division I collegiate football athletes
  Interventions: Other: Education
- CDC Video (Active Comparator): CDC-Vi is an online learning module developed by the CDC and the National Federation of State High School Associations Learning Center. Learners progress through the curriculum sequentially completing each unit before proceeding to the next. The primary narrator of CDC-Vi is Dr. Mick Koester, Chair of the NFHS Sports Medicine Advisory Committee
  Interventions: Other: Education
- CDC Written (Active Comparator): CDC-Wr consists of educational PDFs available for download from the CDC website, as part of the CDC's "Heads Up" brain injury awareness initiative. The PDFs used for the CDC-Wr condition were specific to high school athlete concussion education
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Education

SUMMARY:
Importance: Concussion underreporting leads to delays in diagnosis and treatment, resulting in prolonged recovery. Athletes' report of concussion symptoms is therefore an important component of risk reduction. Numerous educational interventions to improve concussion knowledge and reporting exist.

Objective: Evaluate the comparative efficacy of three concussion education programs in improving concussion-reporting intention.

Design: Randomized clinical trial conducted from August 2018 to October 2018, with assessment before, immediately after, and one-month after educational intervention.

ELIGIBILITY:
Inclusion:

* Athletes from three high school football teams in California.
* In attendance for practice on both study dates
* Provided signed assent and parental consent.

Exclusion:

* Did not complete more than 50% of the questionnaire.

Ages: 14 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — American football players
Enrollment: 118 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Improvement in concussion reporting intention among athletes | 1 month
  All primary and secondary outcomes, besides those related to concussion knowledge, were assessed based on athlete responses, on a 10-point Likert type scale ranging from 1=strongly disagree to 10=strongly agree, to specific questions related to that domain. A composite measure for each outcome was created by summing athletes' responses and dividing by the number of questions asked, resulting in outcomes scaled from 1 to 10.
  A composite measure created based on the inverse of athlete responses to five questions about their concussion-reporting intention (i.e., whether they would continue playing with a concussion during "the beginning of the season," "a practice," "the middle of the season," "during a championship game," and "at the end of the season").

SECONDARY OUTCOMES:
Improvement in concussion knowledge among athletes | 1 month
  Athletes answered 23 True/False questions to assess their concussion knowledge modified from previously utilized concussion educational assessments (Rosenbaum et al., 2010). A composite measure of athlete concussion knowledge was created by summing athletes' correct responses and dividing by the number of questions asked.
  Rosenbaum AM, Arnett PA. The development of a survey to examine knowledge about and attitudes toward concussion in high-school students. J Clin Exp Neuropsychol. 2010;32(1):44-55. doi:10.1080/13803390902806535
Improvement in concussion attitudes among athletes | 1 month
  All primary and secondary outcomes, besides those related to concussion knowledge, were assessed based on athlete responses, on a 10-point Likert type scale ranging from 1=strongly disagree to 10=strongly agree, to specific questions related to that domain. A composite measure for each outcome was created by summing athletes' responses and dividing by the number of questions asked, resulting in outcomes scaled from 1 to 10.
  A composite measure created based on athlete responses to six questions about their attitudes towards concussion reporting (i.e., the extent to which an athlete who reports a concussion would be "better off in the long run," "back on the field much faster," "proud even if teammates call me weak," "better off avoiding participation with signs and symptoms of a concussion," not "better off hiding symptoms from a doctor to not stay out as long," and not "better off toughing it out because concussions are just another injury").
Improvement in concussion perceived normative beliefs among athletes | 1 month
  All primary and secondary outcomes, besides those related to concussion knowledge, were assessed based on athlete responses, on a 10-point Likert type scale ranging from 1=strongly disagree to 10=strongly agree, to specific questions related to that domain. A composite measure for each outcome was created by summing athletes' responses and dividing by the number of questions asked, resulting in outcomes scaled from 1 to 10.
  A composite measure created based on athlete responses to two questions assessing perceived reporting norms (i.e., the extent to which the athlete worried "my teammates would think less of me" if he reported a concussion, or needed to "hide my symptoms from my coach").
Improvement in concussion perceived behavioral control among athletes | 1 month
  All primary and secondary outcomes, besides those related to concussion knowledge, were assessed based on athlete responses, on a 10-point Likert type scale ranging from 1=strongly disagree to 10=strongly agree, to specific questions related to that domain. A composite measure for each outcome was created by summing athletes' responses and dividing by the number of questions asked, resulting in outcomes scaled from 1 to 10.
  A composite measure created based on athlete responses to six questions about their perceived ability and confidence with concussion reporting (i.e., confidence in my ability "to report a concussion," "to help my teammate report a concussion," "to report symptoms of a concussion," "to help my teammate report symptoms of a concussion," "to report symptoms of a concussion, even if I don't think they're that bad," and "to help my teammate report symptoms of a concussion, even if I don't think they're that bad").

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Via contact with study PI, and pending approval of IRB
Supporting Information: Study Protocol